CLINICAL TRIAL: NCT04709653
Title: The Effect of Occupation-Based Nursing Program Applied to Pediatric Oncology Patients on Chemotherapy-Related Symptoms and Satisfaction
Brief Title: The Effect of Occupation-Based Nursing Program Applied to Pediatric Oncology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sule ŞENOL, Research assisstant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Akdeniz Unv
Record Dates: First submitted 2020-11-19; First posted 2021-01-14 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Pediatric Cancer
Keywords: Child; Cancer; Chemotherapy; Occupation; Nursing
MeSH Terms: conditions — Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This was pretest-posttest design, randomized controlled trial.
Masking Description: The control and intervention group will be formed by randomization. The intervention and control group will be defined as group 1 and group 2 for statistical analysis. Data analysis will be evaluated and reported by the statistician. Also the statistician will be blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Occupation-based nursing program
  Interventions: Other: Occupation-based nursing program
- Control Group (Experimental): Routine nursing care
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Occupation-based nursing program — First Session (Rug Weaving Activity): The child and the caregiver will be informed about the purpose and process of the research. The researcher will show in detail how to use rug weaving materials. Rug weaving activity will be started with the child. At the end of the 30-minute practice, the second session with the child will be planned and the session will be ended.
  Second Session (Rug Weaving Event Continues). Third Session (Rug Weaving Activity Continues): Rug weaving activity will be completed and the session will be ended by planning the fourth session with the child.
  Fourth Session (Origami Activity): A figure will be made with origami with the child. The child will be given support to make another figure. The fifth session hour will be planned with the child and the session will be ended.
  Fifth Session (Shape Making Activity with Chenille): A shape will be created with the child with chenille.
  Arms: Intervention Group
Other: Control Group — Routine nursing care
  Arms: Control Group

SUMMARY:
Nurses can include the child in their occupational activities by using the therapeutic communication techniques they have learned during their education. However, there is no occupation-based nursing program that is routinely implemented for children in pediatric clinics. Therefore, the aim of this study is to investigate the effect of occupation-based nursing program on increasing child satisfaction as well as reducing the symptoms of chemotherapy in pediatric oncology patients.

DETAILED DESCRIPTION:
Stressful processes that pediatric oncology patients may be exposed to in the hospital can have a negative effect on the child's anxiety, decrease in activities, and consequently recovery and participation in hospital care. These processes are very difficult for school children as well as for all children. Hospitalization becomes a limiting factor for the school-age child in this period when he is open to mental and physical development, and he starts to attach more importance to socialization and independence. In addition, problems such as painful diagnosis and treatment procedures, side effects of chemotherapy drugs, and insufficient activity support in the hospital may cause the child to stay away from activities. For these reasons, pediatric oncology patients spend their time in their rooms during chemotherapy treatments. With non-pharmacological approaches that can be applied to pediatric oncology patients, chemotherapy-induced symptoms such as fatigue, pain, anxiety and nausea can be reduced, as well as helping to spend the time in the hospital more enjoyable and active. In the studies conducted, it is stated that these approaches are mostly distracting methods. In this context, the use of distraction methods in nursing care is a valuable aspect of care. In our country, randomized controlled studies in which nurses use non-pharmacological methods are quite limited. With the increase of these studies, the use of effective non-pharmacological methods for pediatric oncology patients will be widespread. This study was planned to examine the effect of occupation-based nursing program (OBaNup) in pediatric oncology patients in reducing the symptoms of chemotherapy and on child satisfaction. In the experimental part of the study; It is planned to conduct a randomized controlled single blind experimental study with 60 pediatric oncology patients, including 30 interventions and 30 controls, who received chemotherapy treatment. It is planned to apply OBaNup to the initiative group for an average of 30 minutes a day for five days. Since there is no routine occupation-based nursing program applied to children in the clinic, it is thought that this study can contribute to both the literature and nursing practices. Therefore, in the planned study; It is predicted that OBaNup applied to pediatric oncology patients can reduce the symptoms of chemotherapy and increase satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 7-12 years old,
* Inpatient treatment in Pediatric Hematology-Oncology service,
* Children who can read and write in Turkish will be included in the study.

Exclusion Criteria:

* Those who have visual or upper extremity impairment,
* Mentally disabled,
* Children in terminal period will not be included in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Change of chemotherapy-induced symptoms | at the baseline, immediately upon the completion of the program (fifth day), seven days after the intervention, and before discharge (14 days after the intervention)
  Measured by Memorial Symptom Assessment Scale (7-12) is used to evaluate the symptoms of chemotherapy.
  The scale is an 8-item scale used to evaluate the symptoms of pain, fatigue, sadness, nausea, itching, anxiety, change in taste, and insomnia experienced in the last two days by 7-12 year old children diagnosed with cancer. Symptoms are rated as 'present' or 'absent'. If symptoms are present, their duration is scored as "short duration (1 point)", "medium duration (2 points)" and "long duration (3 points)". The severity of the symptom is scored as "slight", "moderate", and "severe" in the same way as duration. The amount of distress caused by the symptom in the child is scored as "not at all (0 points)", "some (1 point), "moderate (2 points)" and "a lot (3 points)". It is 12. As the score obtained from the scale increases, it indicates that the negative effects of the symptom on the child increase.
Change of psychosocial symptoms for hospitalized children | at the baseline, immediately upon the completion of the program (fifth day), seven days after the intervention, and before discharge (14 days after the intervention)
  Measured by Psychosocial Symptoms Diagnostic Scale for Hospitalized Children The scale developed to diagnose psychosocial symptoms for hospitalized children aged 6-12. Each statement in the 3-point Likert-type scale consisting of 24 items, which can be filled by the practitioner, was evaluated as "never", "sometimes" and "often" and scored as 0, 1 and 2, respectively. The highest score to be obtained from the scale is "48" and the lowest score is "0". A high score on the scale indicates that the child hospitalized in the clinic has psychosocial problems.
Change in satisfaction for hospitalized children | at the baseline, immediately upon the completion of the program (fifth day), seven days after the intervention, and before discharge (14 days after the intervention)
  Measured by Child Satisfaction Form In the form prepared by the researchers in line with the literature, there are 10 questions to evaluate the satisfaction of the pediatric oncology patient. The form is in a five-point Likert type with the answers "I totally agree", "I somewhat agree", "I am undecided", "I do not agree" and "I do not agree at all". The minimum score that can be obtained from the form is 10 and the maximum score is 50. An increase in the scale score indicates that the child's satisfaction increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Şule Şenol, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohammadi A, Mehraban AH, Damavandi SA. Effect of Play-based Occupational Therapy on Symptoms of Hospitalized Children with Cancer: A Single-subject Study. Asia Pac J Oncol Nurs. 2017 Apr-Jun;4(2):168-172. doi: 10.4103/apjon.apjon_13_17. PMID 28503651